CLINICAL TRIAL: NCT00914953
Title: Oxytocin and Social Behavior Over the Lifespan: Interventional Study
Brief Title: Oxytocin and Social Behavior Over the Lifespan
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Responsible Party: Principal Investigator, Paul J. Zak, Professor, Claremont Graduate University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: CNS-R21AG029871; NIH Grant 1R21AG029871-01A2
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Social Activity
Keywords: social isolation; cooperative behavior; depression; loneliness; happiness; empathy
MeSH Terms: conditions — Social Isolation; Cooperative Behavior; Depression | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxytocin (Experimental)
  Interventions: Drug: oxytocin (Pitocin)

INTERVENTIONS:
Drug: oxytocin (Pitocin) — 40 IU OT intranasally (IN) once-daily for 10 consecutive days

SUMMARY:
This study will investigate if intranasal oxytocin (a hormone naturally produced in the body) promotes motivation for, and engagement in, social activities in older adults.

DETAILED DESCRIPTION:
Using a double-blind and placebo controlled design, this study seeks to determine if a short course of exogenous oxytocin (OT) will induce changes in social activities in residentially housed older adults (OAs) during a 10-day treatment period, and after it ends. Because OT is associated with peri-reproductive behaviors, OT release in OAs is expected to be attenuated relative to younger adults. If OT release is low in OAs as we hypothesize, augmenting OT may increase their desire for social interactions, increase the frequency of participation in social activities and augment the number of and quality of social ties, thereby providing protection against disease, early death, cognitive decline, and depression. Research in rodents suggests that social interactions themselves may change chronic OT levels (Carter & Keverne, 2002; Carter & Altemus, 1997), in a positive feedback loop. In order to demonstrate OT as the causal mechanism, we propose to infuse oxytocin and then track the desire for, quantity of, and quality of social activities.

ELIGIBILITY:
Inclusion Criteria:

* residentially housed
* English fluency

Exclusion Criteria:

* non ambulatory
* severe psychiatric problems presently or in the recent past
* severe medical problems (e.g., cancer, diabetes, advanced heart disease)
* irregular heart beat
* treatment using psychoactive medications (other than antiepileptics, mood stabilizers, or Ambien)
* inability to adequately communicate with the research team
* treatment with an experimental drug
* excessive fatigue suggesting hypothyroidism

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
confirm increased social activities in treatment condition compared to control condition via self-report. | 30 days

SECONDARY OUTCOMES:
Evidence of greater psychological health for treatment condition as compared to control condition. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Linda Valley Villa, Loma Linda, California, United States